CLINICAL TRIAL: NCT07120386
Title: Instillation vs Traditional Negative Pressure Wound Therapy: A Pilot Randomized Controlled Trial for Necrotizing Soft Tissue Infections (NPWTi-NSTI Trial)
Brief Title: Irrigating vs Traditional Negative Pressure Wound Therapy to Treat Necrotizing Soft Tissue Infections
Acronym: NPWT-NSTI
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: HealthPartners Institute (Other)
Collaborators: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: A24-205; 0002758892 (Other Grant/Funding Number: University of Minnesota Translational Center for Resuscitative Trauma Care)
Record Dates: First submitted 2025-07-25; First posted 2025-08-13 (Actual); Last update posted 2025-09-17 (Actual); Status verified 2025-09

CONDITIONS: Necrotizing Soft Tissue Infections
Keywords: Negative pressure wound therapy; NPWT; NPWTi
MeSH Terms: interventions — Negative-Pressure Wound Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Negative Pressure Wound Therapy (Active Comparator): Patients in this arm will receive traditional Negative Pressure Wound Therapy (NPWT)
  Interventions: Device: Negative Pressure Wound Therapy
- Negative Pressure Wound Therapy with Instillation (Experimental): Patients in this arm will receive Negative Pressure Wound Therapy with Instillation of a hypochlorous acid solution (NPWTi)
  Interventions: Device: Negative Pressure Wound Therapy with Instillation

INTERVENTIONS:
Device: Negative Pressure Wound Therapy — NPWT creates a vacuum seal over your wound to promote healing
  Other Names: NPWT
  Arms: Negative Pressure Wound Therapy
Device: Negative Pressure Wound Therapy with Instillation — NPWTi creates a vacuum seal over your wound and infuses the wound with hypochlorous acid (medical grade dilute bleach) to clean it.
  Other Names: NPWTi
  Arms: Negative Pressure Wound Therapy with Instillation

SUMMARY:
Necrotizing Soft Tissue Infections (NSTIs) are rapidly progressing infections that have a high morbidity and mortality, with the greatest morbidity related to managing the large wounds required to treat these patients. Initial treatment requires wide surgical removal of infected tissue and optimal management is essential to reducing morbidity in these patients. Negative pressure wound therapy (NPWT) is a widely used technology that has revolutionized wound management. NPWT is utilized across the spectrum of acute wounds, including routine postoperative incision management, traumatic wounds, and wounds related to surgical debridement of NSTIs which are frequently some of the most complicated of wounds encountered. Most NSTI cases at Regions Hospital currently utilize negative pressure wound therapy with instillation (NPWTi) where the wound is irrigated to clean out debris. Currently, there is a paucity of data comparing traditional NPWT and NPWTi and the choice of which device to use is left to surgeon discretion. This study is a first step at identifying the effects of NPWTi compared to NPWT alone on the care of NSTI patients. If the theoretical benefits of NPWTi over NPWT translate to practice, those treated with NPWTi would be expected to have a reduced rate of hospital readmission after their index hospitalization in addition to shorter time to definitive closure/coverage. This is a pilot study to assess the feasibility of enrolling patients with NSTIs in a randomized controlled trial to assess outcomes between the two devices.

ELIGIBILITY:
Inclusion Criteria:

* Clinical suspicion for Necrotizing Soft Tissue Infection (NSTI) necessitating emergent operative intervention
* Age >/=18 years old
* Planned application of a negative pressure wound dressing

Exclusion Criteria:

* Patients who have a wound that does not allow for a wound vac
* Patients receiving acute treatment for a NSTI at another institution
* Incarcerated patients
* Patients who do not survive to wound closure/coverage
* Patients <18 years old

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-08-01 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Unplanned hospital readmission | Within 30 days of discharge
  Did the patient have an unplanned readmission to the hospital (Y/N) within 30 days of discharge
Rate of healing | First operation and last operation
  Time from index debridement to final coverage in days

OTHER OUTCOMES:
Number of operative interventions | Through hospital discharge, median of 9 days
  Number of times the patient required an operation related to their NSTI during their hospital stay
Unplanned vac change | Through hospital discharge, median of 9 days
  Number of unplanned times the vacuum dressing had to be changed during their hospital stay
Total vac changes | Through hospital discharge, median of 9 days
  Total number of times the vacuum dressing was changed (planned + unplanned) during their hospital stay
Bleeding | Through hospital discharge, median of 9 days
  Bleeding at wound vac site (Y/N). During hospital stay
Infection | Through hospital discharge, median of 9 days
  New infection at wound vac site (Y/N). During hospital stay
Hospital length of stay | At hospital discharge, median of 9 days
  Number of days spent in Hospital
Intensive Care Unit length of stay | At hospital discharge, median of 9 days
  Number of days spent in the Intensive Care Unit
Floor length of stay | At hospital discharge, median of 9 days
  Number of days spent inpatient in the hospital
Skilled Nursing Facility days | Up to 6 months after admission to skilled nursing facility
  Number of days spent in a skilled nursing facility
Discharge disposition | At hospital discharge, median of 9 days
  "Where was the patient discharged: ""1=Discharged/Transferred to a short-term general hospital for inpatient care 2=Discharged/Transferred to an Intermediate Care Facility (ICF) 3=Discharged/Transferred to home under care of organized home health service 4=Left against medical advice or discontinued care 5=Deceased/Expired 6=Discharged to home or self-care (routine discharge) 7=Discharged/Transferred to Skilled Nursing Facility (SNF) 8=Discharged/Transferred to hospice care 9=Discharged/Transferred to court/law enforcement. 10=Discharged/Transferred to inpatient rehab or designated unit 11=Discharged/Transferred to Long Term Care Hospital (LTCH) 12=Discharged/Transferred to a psychiatric hospital or psychiatric distinct part unit of a hospital 13=Discharged/Transferred to another type of institution not defined elsewhere"""

CONTACTS AND LOCATIONS:
Overall Officials: Brian S Myer, MD, Principal Investigator — Regions Hospital
Locations (1):
- Regions Hospital, Saint Paul, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No